CLINICAL TRIAL: NCT06978205
Title: Effect of Urethral Balloon Dilatation on Urinary Retention After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYLL-202503-011-1
Record Dates: First submitted 2025-05-05; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries (SCI); Urinary Bladder, Neurogenic; Urinary Retention
Keywords: Spinal Cord Injuries; neurogenic bladder; urinary retention; Urethral balloon dilation; zelen design; Randomized controlled clinical trial
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Retention | interventions — Intermittent Urethral Catheterization; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rehabilitation treatment. (Active Comparator): Conventional rehabilitation treatment methods include intermittent catheterization, acupuncture and pelvic floor function training. Intermittent catheterization is based on the results of urodynamic examination to develop a personalized drinking plan and the number of catheterization, and the number of catheterization is selected according to the amount of residual urine. Acupuncture treatment improves the patient's urinary function by acupuncture on the lower abdomen and lumbosacral acupoints once a day, 5 days a week, for a total of 1-2 weeks. The pelvic floor therapist assesses the patient's pelvic floor muscle condition and guides the patient to perform effective pelvic floor muscle contractions and relaxations.
  Interventions: Device: intermittent catheterization; Device: Acupuncture treatment; Behavioral: Pelvic floor function training
- Urethral Balloon Dilation (Experimental): 1.A 14-Fr urethral catheter will be prefilled with sterile saline to check for balloon integrity. If intact, the saline will be completely withdrawn. 2.Ultrasound imaging will be used to precisely locate the external urethral sphincter. 3.The catheter will be fully lubricated and gently inserted into the urethra. 4.Under real-time ultrasound guidance, 2-4 mL of sterile saline will be gradually injected into the balloon to expand the external urethral sphincter. 5.Patients will be instructed to attempt urination during the procedure, and changes in voiding patterns will be observed. This procedure will be performed three times per participant. The expansion volume will increase by 0.5-1 mL per session, depending on urethral outlet resistance (urodynamic results) and degree of urethral narrowing (ultrasound assessment）Each session lasts 5 minutes. Strict aseptic techniques will be followed.
  Interventions: Device: Urethral Balloon Dilation; Device: intermittent catheterization; Device: Acupuncture treatment; Behavioral: Pelvic floor function training

INTERVENTIONS:
Device: Urethral Balloon Dilation — Urethral balloon dilation + conventional rehabilitation therapy. 1.A 14-Fr urethral catheter will be prefilled with sterile saline to check for balloon integrity. If intact, the saline will be completely withdrawn. 2.Ultrasound imaging will be used to precisely locate the external urethral sphincter. 3.The catheter will be fully lubricated and gently inserted into the urethra. 4.Under real-time ultrasound guidance, 2-4 mL of sterile saline will be gradually injected into the balloon to expand the external urethral sphincter. 5.Patients will be instructed to attempt urination during the procedure, and changes in voiding patterns will be observed. This procedure will be performed three times per participant. The expansion volume will increase by 0.5-1 mL per session, depending on urethral outlet resistance (urodynamic results) and degree of urethral narrowing (ultrasound assessment）Each session lasts 5 minutes. Strict aseptic techniques will be followed.
  Arms: Urethral Balloon Dilation
Device: intermittent catheterization — Intermittent catheterization is based on the results of urodynamic examination to develop a personalized drinking plan and the number of catheterization, and the number of catheterization is selected according to the amount of residual urine.
Device: Acupuncture treatment — Acupuncture treatment improves the patient's urinary function by acupuncture on the lower abdomen and lumbosacral acupoints.
Behavioral: Pelvic floor function training — The pelvic floor therapist assesses the patient's pelvic floor muscle condition and guides the patient to perform effective pelvic floor muscle contractions and relaxations.

SUMMARY:
Trial Objectives: This clinical trial aims to explore whether ultrasound - guided urethral balloon dilation can effectively improve the micturition function of patients with urinary retention after spinal cord injury, and to evaluate the safety of this treatment method. The main questions it attempts to answer are:

Can ultrasound - guided urethral balloon dilation reduce the residual urine volume and improve the quality of life of patients with urinary retention after spinal cord injury? Trial Design: Researchers will compare the group receiving ultrasound - guided urethral balloon dilation combined with conventional rehabilitation therapy (the experimental group) with the group receiving only conventional rehabilitation therapy (the control group) to determine the therapeutic effect of ultrasound - guided urethral balloon dilation on urinary retention after spinal cord injury.

Tasks for Participants:

Participants in the experimental group will receive ultrasound - guided urethral balloon dilation and cooperate with conventional rehabilitation therapy (including acupuncture therapy, pelvic floor biofeedback electrical stimulation, and pelvic floor function training). Participants in the control group will receive only conventional rehabilitation therapy for a period of 1 - 2 weeks.

During the intervention, patients are required to strictly record a micturition diary under the guidance of researchers or medical staff. The diary should cover details such as daily spontaneous urine output, daily catheterized urine output, daily urine leakage volume, and daily frequency of catheterization.

Residual urine volume will be detected every day for three days before the intervention and three days after the intervention.

DETAILED DESCRIPTION:
Standard Rehabilitation Treatment (Control Group)：Participants in the control group will receive conventional rehabilitation therapy: Pelvic floor muscle training and Biofeedback electrical stimulation.

Urethral Balloon Dilation (Intervention Group)：Participants in the intervention group will receive urethral balloon dilation in addition to standard rehabilitation therapy. The specific procedures are as follows:

1. A 14-Fr urethral catheter will be prefilled with sterile saline to check for balloon integrity. If intact, the saline will be completely withdrawn.
2. Ultrasound imaging will be used to precisely locate the external urethral sphincter.
3. The catheter will be fully lubricated and gently inserted into the urethra.
4. Under real-time ultrasound guidance, 2-3.5 mL of sterile saline will be gradually injected into the balloon to expand the external urethral sphincter.
5. Patients will be instructed to attempt urination during the procedure, and changes in voiding patterns will be observed.
6. After treatment, the balloon will be fully deflated, and the catheter will be carefully removed.

This procedure will be performed three times per participant. The expansion volume will increase by 0.5-1 mL per session, depending on urethral outlet resistance (urodynamic results) and degree of urethral narrowing (ultrasound assessment). Each session lasts 5 minutes. Strict aseptic techniques will be followed. The procedure will be conducted by experienced physicians under ultrasound guidance to ensure maximum safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80 years old
2. There is a confirmed diagnosis report of CT or MRI imaging, with the first diagnosis being spinal cord injury (complete or incomplete), which conforms to the International Classification of Spinal Cord Injury Neurology published by the American Spinal Injury Association (ASIA) in 2013
3. The spinal shock period has passed, and consciousness is clear with stable vital signs
4. In line with the diagnostic criteria of urinary retention and in combination with clinical practice: the patient can urinate autonomously before spinal cord injury, which is confirmed as spinal cord injury by clinical examination. It is manifested as retention of urine after spinal cord injury, swelling of lower abdomen, filling of bladder, dullness on percussion, residual urine volume of bladder B ultrasonic examination is more than 300ml, which shows that urination is laborious
5. Urodynamic examination shows maximum urethral pressure greater than 50cmH2O
6. No tumors or benign prostatic hyperplasia were found
7. Patients who have had their indwelling urinary catheter removed
8. Voluntary participation in research and signing of informed consent form

Exclusion Criteria:

1. Patients with severe heart, brain, lung and other important organ diseases or mental and cognitive disorders
2. Individuals with disrupted water electrolyte and acid-base balance
3. There are serious kidney diseases, bladder fistula surgery, anterior urethral sphincterotomy and other diseases
4. There is a urinary system infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Residual urine volume | Before treatment and three consecutive days after treatment
  Use a bladder capacity measuring instrument (model HD5, produced by Liaoning Hande Technology Co., Ltd.) to perform ultrasound testing on patients after urination and record residual urine volume.
Voiding Diary | Before treatment and three consecutive days after treatment
  Under the supervision of researchers and medical staff, patients were instructed to keep a urinary diary during hospitalization (including catheterization time, spontaneous displacement, catheterization volume, and catheterization frequency)

SECONDARY OUTCOMES:
Short-Form Health Survey-Qualiveen (SF-Qualiveen) | Before treatment and on the third day after treatment
  For the assessment of patients' quality of life, the SF Qualiveen Quality of Life Scale score was used.The scale includes 4 dimensions and 8 items of annoyance (items 1~2), restriction (items 3~4), fear (items 5~6), and feeling (items 7~8). Each item was scored by Likert 5 grades, in which item 3 was assigned a score of "never", "rarely", "sometimes", "often" and "always", and the rest of the items were assigned 0~4 points according to "none", "a little", "moderate", "quite severe" and "extremely severe", the score of each dimension was the mean of each item within the dimension, and the score of the scale was the average score of each dimension, with a total score of 0~4 points, the lower the score, the better the quality of life of patients.
Neurogenic Bladder Symptom Score (NBSS) | Before treatment and on the third day after treatment
  The NBSS Neurogenic Bladder Symptom Rating Scale was used to score the patient's urinary symptoms.The NBSS scale consists of 24 items assessing three key dimensions: urinary incontinence (8 items, 0-29 points), bladder storage and voiding function (7 items, 0-22 points), urinary tract complications (7 items, 0-23 points). Additionally, two non-scoring items assess bladder management methods and overall quality of life. Each item is scored from 0 to 3 or 0 to 4, with higher scores indicating more severe bladder symptoms.
Core Lower Urinary Tract Symptom Rating Scale | Before treatment and on the third day after treatment
  CLSS will be used to evaluate lower urinary tract symptoms before and after treatment. The total score ranges from 0 to 30: 0 points = No symptoms, 1 point = Rare symptoms, 2 points = Occasional symptoms, 3 points = Frequent symptoms, Lower CLSS scores indicate greater symptom improvement following treatment
Hospital Anxiety and Depression Scale (HADS) | Before treatment and on the third day after treatment
  The HADS was developed by Zigmond AS and Snaith RP in 1983 for screening anxiety and depression in hospitalized patients[36]. The scale consists of 14 items, divided into: 7 items for depression assessment, 7 items for anxiety assessment, The Chinese version of HADS has demonstrated strong reliability and validity, making it an effective tool for assessing psychological well-being in clinical settings

CONTACTS AND LOCATIONS:
Locations (1):
- Hui Wei, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No